CLINICAL TRIAL: NCT04476654
Title: Improving Uptake of Genetic Cancer Risk Assessment in African American Women- Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-19-15167; HM20016234 (Other: VCU IRB); NCI-2019-04689 (Other: CTRP); R21CA236496 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-07-20 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: genetic counseling and testing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fact Sheet Arm (No Intervention): Komen print materials about genetic counseling and testing will be given to women.
- YouTube Video Arm (Active Comparator): Participants in this arm will receive the culturally tailored video either via a Youtube link or a DVD.
  Interventions: Behavioral: YouTube Video Arm

INTERVENTIONS:
Behavioral: YouTube Video Arm — Participants (n=25) will watch a 20 minute YouTube video that will describe the genetic counseling and testing process and risk/benefit information in a culturally relevant format. Participants will complete pre and post assessments. After the session, participants interested in pursuing genetic counseling and testing services will be referred to a patient navigator who will navigate participants to identified no cost or low cost services.
  Arms: YouTube Video Arm

SUMMARY:
Genetic counseling and testing (GCT) provides invaluable information for women who are at-risk of hereditary breast and/or ovarian cancer (HBOC). Black women underutilize GCT compared to White women. This study will conduct a RCT to test the efficacy of a culturally-tailored theory-based video intervention aimed to address key psychosocial factors (emotions, ambivalence) to improve uptake of genetic counseling in Black women at increased risk of HBOC. Findings from this study may offer an opportunity to engage at-risk Black women regarding genetic counseling through a multi-center trial and ultimately address the disparity in genetic counseling uptake that exists between Black and White women.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most frequently diagnosed cancer in African American women (hereafter referred to as "Black") and their cancer mortality is higher than other racial/ethnic groups in the United States (US). Compared to non-Hispanic Whites, Black women are diagnosed younger and with more advanced breast cancer. When diagnosed with BC, Black women present more often with triple-negative breast cancer (TNBC) an aggressive disease defined by the absence of estrogen and progesterone receptors, and human epidermal growth factor (HER)-2 expression. TNBC has been associated with pathogenic BRCA1 variants. Racial disparities also exist for women with ovarian cancer, the most lethal of the gynecologic cancers. Among women with advanced ovarian cancers up to 21% are associated with inherited pathogenic mutations the most common of which is BRCA1. Women who carry a pathogenic BRCA variant (PV) have a lifetime breast cancer risk of 55-70% and a lifetime ovarian cancer risk of up to 44%. The National Comprehensive Cancer Network (NCCN) recommends referral for Hereditary Breast and Ovarian Cancer (HBOC) genetic counseling and testing (GCT) for women at risk of carrying a BRCA PV. GCT provides women with information needed to make informed decisions to reduce their cancer risk, yet Black women are less likely to use GCT than whites. There is a dearth of interventions to address this issue and produced results are mixed and modest. Awareness of a positive result can inform treatment decisions for cancer patients and risk management in survivors or women unaffected with cancer.

Reasons for the lower uptake of GCT in Black women are multi-factorial and include access, knowledge, psycho-social factors, and may vary by cancer status (affected versus unaffected). There are substantial scientific gaps regarding effective interventions to address the sub-optimal uptake of GCT in Black women. To be effective, GCT interventions should be anchored within the needs and cultural values of their audience. While improving knowledge about GCT and one's individual risks is important, interventions that only address knowledge may not enhance uptake, as risk information evokes emotional reactions that are often stronger predictors of behaviors than cognitive factors.

Notably, this team has identified factors that contribute to Black women's uptake of GCT. In preliminary studies, researchers found that self-efficacy in making decisions about GCT and medical mistrust were associated with GCT uptake. Low knowledge among Black BC survivors at risk of HBOC has also been found. Anticipated negative emotions to GCT have been associated with lower uptake. Similar studies suggest that Black women report emotions related to fear of being singled out, and the fear of being hopeless. Because most interventions have focused solely on knowledge or access, the proposed study makes a considerable shift in the field by additionally targeting emotions, ambivalence, and developing a media-based risk communication tool.

Guided by two evidenced-based theories and preliminary data, this will be a two-phased mixed methods study. In Phase I (months 1-7), formative research and preliminary data will be used to develop the script for the GCT video. The script will be reviewed by GCT experts (n=4) and piloted in two focus groups (n=16) followed by a staged reading to make final refinements. In Phase II (months 8-24), a two-arm randomized trial (RCT) to compare GCT uptake and psycho-social outcomes between 50 at-risk Black women receiving printed Susan G. Komen developed GCT literature (control group) (n=25) or a tailored YouTube video intervention (n=25) will be conducted . All women will be referred to an appointment scheduler who will assist them with making an appointment with a genetic counselor. Participants will complete a baseline survey and follow-up assessment. The primary outcome will be genetic counseling uptake and receipt testing at 3-months will be explored. Specific aims are to:

Aim 1. Develop a YouTube video using a formative data for Black women at risk for HBOC.

Aim 2. Evaluate the efficacy of the intervention by comparing outcomes between women in the YouTube intervention arm vs. control group arm. H.2.1. Women in the intervention group (vs control group) will have higher genetic counseling uptake. H.2.2. Women in the intervention group (vs control group) will report higher knowledge, higher self-efficacy, higher endorsement of positive attitudes, and positive anticipated emotions about GCT. H.2.3. Most women (≥75%) will be satisfied with the experimental intervention.

Enhancing GCT in at-risk populations is a national priority. Given trends towards panel testing and other genomic advances, there is potential for existing disparities to widen. Findings will inform new strategies for behavioral interventions for Black women and a larger trial. If successful, the intervention could be easily disseminated broadening its reach to affected and unaffected women.

This study meets the Healthy People 2020 goals to enhance GRCA in at-risk populations, and the national priorities to increase diversity in genetics research participation and incorporate emotions into cancer research. Findings will inform new strategies for behavioral interventions targeting African-Americans in a larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must be at high risk for hereditary breast or ovarian cancer
* Must identify as Black/African American
* Must be a woman
* Referred to a genetic counselor for the purpose of being high risk of carrying a hereditary breast and/or ovarian cancer mutation

Genetic Counselors:

* Must be at least 18 years of age
* Must be qualified
* Must be approved by the PI

Exclusion Criteria:

* Under the age of 18
* Race other than Black/African American
* Do not gave a high risk for hereditary breast or ovarian cancer

Genetic Counselors:

* Under 18
* Not qualified
* Not approved by the PI

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Sheppard, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trained clinical coordinators recruited participants, administered surveys and abstracted information on genetic counseling and testing from participant medical records
Pre-assignment Details: The clinical research assistants consented interested patients . Following consent, women completed a baseline survey. Next, women were randomized into study arms.
Period: Overall Study
Arm/Group | Fact Sheet Arm | YouTube Video Arm
Started | 29 | 28
Completed | 26 | 26
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fact Sheet Arm | YouTube Video Arm | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.24 (16.91) | 49.50 (13.38) | 48.35 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 29 | 28 | 57
Genetic Counseling Knowledge [Mean (Standard Deviation); unit: units on a scale] | 7.69 (1.75) | 7.50 (1.45) | 7.60 (1.60)
Self-Efficacy to Screen [Mean (Standard Deviation); unit: units on a scale] | 14.38 (1.21) | 14.29 (2.32) | 14.33 (1.83)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Genetic Counseling and Testing Uptake.
Description: Our primary outcome will be for participants to receive genetic testing and counseling.Investigators will be able to see if participant has scheduled a genetic testing appointment within the VCU Health appointment system.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fact Sheet Arm | YouTube Video Arm
Number analyzed (Participants) | 29 | 28
Participants
  Counseling | 18 | 15
  Testing | 7 | 12

2. Secondary Outcome: Knowledge Scale - Genetic Counseling and Testing Knowledge .
Description: The investigators measured general knowledge about hereditary breast and ovarian cancer. GCT knowledge was ascertained using a 13 item scale developed by Erblich et al.'s (2005). Example items included "have you ever heard about genetic counseling for BRCA 1 and 2?"" and have yes/no or true/false options. Scores across the 13 item Knowledge scale were summed with a range of ( 0-13) where higher values indicated higher knowledge.
Time Frame: Baseline was collected up to 48 hours from the start of the intervention and the follow-up was assessed within 48 hours post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fact Sheet Arm | YouTube Video Arm
Number analyzed (Participants) | 26 | 26
score on a scale
  Follow-up | 7.79 (1.90) | 8.11 (1.55)
  Baseline | 7.69 (1.75) | 7.50 (1.45)

3. Secondary Outcome: Self-efficacy Scale
Description: The investigators measured participants self-efficacy in genetic counseling services.Self-efficacy was measured with 3 items on a 5-point likert-scale, with questions that was developed for this study. Example items include "how confident are you that you can cope with your risk of developing cancer?". Response options are on a 5-point likert scale ranging from not at all confident (1) and very confident (5). Scores across the 3- item scale were summed with a range of (3-15) where higher scores indicated higher self efficacy.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fact Sheet Arm | YouTube Video Arm
Number analyzed (Participants) | 26 | 26
score on a scale
  Follow-up | 14.76 (0.91) | 14.21 (2.02)
  Baseline | 14.38 (1.21) | 14.29 (2.32)

ADVERSE EVENTS:
Time Frame: N/A no Adverse Event (AE) data was collected per the protocol
Description: N/a no AE data was collected per the protocol
Arm/Group | Fact Sheet Arm | YouTube Video Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT04476654/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT04476654/SAP_002.pdf
  • Informed Consent Form (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04476654/ICF_000.pdf